CLINICAL TRIAL: NCT01296438
Title: A Randomised Trial Investigating the Pharmacokinetic Properties of NN1218 in Subjects With Type 1 Diabetes
Brief Title: A Trial Investigating the Pharmacokinetic Properties of NN1218 in Subjects With Diabetes Mellitus, Type 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3872; 2010-022222-33 (EudraCT Number); U1111-1118-6955 (Other: WHO)
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence 1 (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- Treatment sequence 2 (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Single dose of 0.2 U/kg body weight faster-acting insulin aspart injected subcutaneously (under the skin) followed by single dose of 0.2 U/kg body weight insulin aspart injected subcutaneously (under the skin)
  Other Names: NN1218
  Arms: Treatment sequence 1
Drug: insulin aspart — Single dose of 0.2 U/kg body weight insulin aspart injected subcutaneously (under the skin) followed by single dose of 0.2 U/kg body weight faster-acting insulin aspart injected subcutaneously (under the skin)
  Arms: Treatment sequence 2

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the pharmacokinetic (the rate at which the body eliminates the trial drug) and pharmacodynamic (the effect of the trial drug on the body) profiles of NN1218 in comparison with insulin aspart.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least 12 months
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion (CSII) for more than 12 months.
* Body Mass Index (BMI) between 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to trial start
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | from 0-1 hour after trial drug administration

SECONDARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | from 0-12 hours after trial drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com